CLINICAL TRIAL: NCT01007136
Title: TDCS-enhanced Stroke Recovery and Cortical Reorganization
Brief Title: Transcranial Direct Current Stimulation (tDCS)-Enhanced Stroke Recovery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding limit reached due to slower then anticipated recruitment.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Timea Hodics, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 092010-231; K23HD050267 (NIH)
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Ischemic Stroke
Keywords: tDCS; stroke; functional MRI; TMS
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Transcranial Direct Current Stimulation; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tDCS and occupational therapy (Experimental): 1 mA electric current will be delivered over the lesioned motor cortex for the first 20 minutes during the one hour physical therapy.
  Interventions: Device: tDCS
- Sham and occupational therapy (Sham Comparator): Electric current will be ramped up and down over the lesioned motor cortex for the first seconds during the one hour physical therapy.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — 1 mA electric current will be delivered over the lesioned motor cortex for the first 20 minutes during the one hour physical therapy.
  Other Names: Transcranial Direct Current Stimulation; Electric stimulation
  Arms: tDCS and occupational therapy
Device: Sham tDCS — Electric current will be ramped up and down over the lesioned motor cortex for the first seconds during the one hour physical therapy.
  Arms: Sham and occupational therapy

SUMMARY:
The purpose is to determine whether application of a non-invasive battery powered device called transcranial direct current stimulation (tDCS) can improve recovery of hand weakness after stroke beyond what is achievable with rehabilitative treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke causing arm weakness within 5-15 days
* no other neurological or psychiatric disease, who are able to perform study tasks

Exclusion Criteria:

* patients younger than 18 or older than 80 years
* patients with more than one disabling stroke
* Patients with bilateral motor impairment
* Patients with poor motivational capacity, history of severe alcohol or drug abuse
* Patients with severe language disturbances, particularly of receptive nature
* Patients with serious cognitive deficits (defined as equivalent to a MMS score of 23 or less)
* Patients with severe uncontrolled medical problems (e.g., seizures, progressive stroke syndromes, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age or others),
* Patients with unstable thyroid disease
* Patients with increased intracranial pressure
* Patients with unstable cardiac arrhythmia
* Patients with contraindication to TMS or tDCS stimulation (pacemaker, an implanted medication pump, a metal plate in the skull, or metal objects inside the eye or skull, patients who had a craniotomy, skin lesions at the site of stimulation)
* Patients who are not available for follow-up at 3 and 12 months
* Pregnancy
* Patients with contraindication to MRI will not participate in MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Hidler J, Hodics T, Xu B, Dobkin B, Cohen LG. MR compatible force sensing system for real-time monitoring of wrist moments during fMRI testing. J Neurosci Methods. 2006 Sep 15;155(2):300-7. doi: 10.1016/j.jneumeth.2006.01.016. Epub 2006 Feb 21. PMID 16490258
- [Background] Hodics TM, Nakatsuka K, Upreti B, Alex A, Smith PS, Pezzullo JC. Wolf Motor Function Test for characterizing moderate to severe hemiparesis in stroke patients. Arch Phys Med Rehabil. 2012 Nov;93(11):1963-7. doi: 10.1016/j.apmr.2012.05.002. Epub 2012 May 10. PMID 22579647
- [Derived] Hodics T, Cohen LG, Pezzullo JC, Kowalske K, Dromerick AW. Barriers to Enrollment in Post-Stroke Brain Stimulation in a Racially and Ethnically Diverse Population. Neurorehabil Neural Repair. 2022 Sep;36(9):596-602. doi: 10.1177/15459683221088861. Epub 2022 Aug 4. PMID 35925037
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: UT SOuthwestern Hospitals, rehabilitation and stroke clinics were screened for eligible stroke patients from 2009 through 2014.
Pre-assignment Details: Enrolled participants were assigned to groups unless they were found to meet one of the exclusion criteria, or withdrew their consent.
Groups:
- fMRI Control Group no Intervention: Healthy volunteers and chronic stroke volunteers were enrolled in the fMRI and TMS component of the study, no intervention was performed.The purpose of this study subgroup was to set up and test the complex MRI and TMS protocol developed for this project.
- tDCS and no Arm Movement: 1 mA electric current was delivered over the lesioned motor cortex for the first 20 minutes during the one hour physical therapy. Same inclusion criteria as the main group except for no UE movement at enrollment.
  tDCS: 1 mA electric current was delivered over the lesioned motor cortex for the first 20 minutes during the one hour physical therapy.
- Sham and no Arm Movement: Sham tDCS: Electric current was ramped up and down over the lesioned motor cortex for the first seconds during the one hour physical therapy.
Period: Overall Study
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | fMRI Control Group no Intervention | tDCS and no Arm Movement | Sham and no Arm Movement
Started | 19 | 17 (One additional subject was excluded prior to randomization due to illicit drug use.) | 15 | 6 | 4
Completed | 15 | 13 | 15 | 6 | 4
Not Completed | 4 | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject who did not meet enrollment criteria was erroneously enrolled and was removed by PI from the study immediately after enrollment, prior to randomization. Therefore the total number of enrolled is one more then randomized.
Groups:
- tDCS and Occupational Therapy: 1 mA electric current was delivered over the lesioned motor cortex for the first 20 minutes during the one hour physical therapy.
  tDCS: 1 mA electric current was delivered over the lesioned motor cortex for the first 20 minutes during the one hour physical therapy.
- Sham and Occupational Therapy; Sham and no Arm Movement: Electric current was ramped up and down over the lesioned motor cortex for the first seconds during the one hour physical therapy.
  Sham tDCS: Electric current was ramped up and down over the lesioned motor cortex for the first seconds during the one hour physical therapy.
- fMRI Control Group no Intervention: Healthy volunteers and chronic stroke volunteers were enrolled in the fMRI and TMS component of the study, no intervention was performed.
- Total: Total of all reporting groups
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | fMRI Control Group no Intervention | tDCS and no Arm Movement | Sham and no Arm Movement | Total
Number analyzed (Participants) | 19 | 17 | 15 | 6 | 4 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 15 | 2 | 3 | 42
  >=65 years | 9 | 5 | 0 | 4 | 1 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.3) | 60.7 (10.3) | 49 (13) | 66 (10) | 63.5 (8.3) | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 9 | 3 | 1 | 32
  Male | 11 | 6 | 6 | 3 | 3 | 29

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Fugl-Meyer
Description: Motor outcome measure for the upper extremity. Scores vary between 0-66, higher values mean better performance.
Time Frame: 2 weeks
Population: All subjects with outcome data at the prespecified follow-up timepoint were included.
  "fMRI Control Group no Intervention" subgroup did not have clinical intervention or clinical outcome measures performed, their data was used for the fMRI and TMS component of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 15 | 13 | 6 | 4
units on a scale | 30.2 (21.2) | 36.8 (22.4) | 8.2 (10.2) | 4.5 (1)

2. Primary Outcome: Upper Extremity Fugl-Meyer
Description: Motor outcome measure for the upper extremity. Scores vary between 0-66, higher values mean better performance.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 10 | 11 | 3 | 1
units on a scale | 32.4 (24.5) | 47.7 (18.7) | 9.7 (9.8) | 4.0 (0.0)

3. Primary Outcome: Upper Extremity Fugl-Meyer
Description: Motor outcome measure for the upper extremity. Scores vary between 0-66, higher values mean better performance.
Time Frame: 1 year after stroke
Population: All subjects with outcome data at the prespecified follow-up timepoint were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 5 | 9 | 0 | 1
units on a scale | 32.6 (29.2) | 56.0 (12.8) |  | 4.0 (0.0)

4. Secondary Outcome: Wolf Motor Function Test
Description: The Wolf Motor Function Test (WMFT) is a quantitative index of upper extremity motor ability determined through the use of timed and functional tasks. The score represents the average speed the subject could perform of the timed motor tasks.
  The score is the average of the scores calculated from "how many times would a person have completed the task, had he or she been performing it continuously for 60 seconds". The score ranges from 0 to no theoretical maximum, with higher numbers meaning faster/ better performance. (See publication Dr. Hodics et al. 2012.)
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 10 | 11 | 2 | 1
units on a scale | 19.7 (19.6) | 30.9 (21.7) | 0.80 (1.12) | 0.79 (0.00)

5. Other Pre Specified Outcome: Visual Analog Pain Scale
Time Frame: during therapy
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mini Mental Status Scale
Description: Mini Mental Status Scale is a test of cognitive function; it includes tests of orientation, attention, memory, language and visual-spatial skills, scored 0-30, the higher scores mean the better performance.
Time Frame: 3 months
Population: fMRI Control Group no Intervention" subgroup did not have clinical intervention or clinical outcome measures performed, their data was used for the fMRI and TMS component of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 10 | 11 | 3 | 1
score on a scale | 24.7 (6.6) | 26.6 (4.8) | 27.3 (3.8) | 30.0 (0.0)

7. Other Pre Specified Outcome: NIHSS
Description: The National Institutes of Health Stroke Scale (NIHSS) provides a quantitative measure of stroke-related neurologic deficit. The NIHSS was originally designed as a research tool to measure baseline data on patients in acute stroke clinical trials. The score ranges 0-42, a score of 0 represents no deficit, lower score is better.
Time Frame: 3 months
Population: All available data from participants was included at the 3 months follow-up. fMRI Control Group no Intervention" subgroup did not have clinical intervention or clinical outcome measures performed, their data was used for the fMRI and TMS component of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 10 | 11 | 2 | 1
units on a scale | 3.50 (3.06) | 1.45 (1.57) | 7.00 (1.00) | 6.00 (0.00)

8. Other Pre Specified Outcome: Beck Depression Inventory
Description: 21-item, self-rated scale that evaluates key symptoms of depression. The minimum score is 0 and maximum score is 63. Higher scores indicate greater symptom severity.
Time Frame: 3 months
Population: All participants with available measurement were included. fMRI Control Group no Intervention" subgroup did not have clinical intervention or clinical outcome measures performed, their data was used for the fMRI and TMS component of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 10 | 11 | 2 | 1
units on a scale | 3.2 (2.9) | 5.0 (4.5) | 5.50 (3.54) | 3.00 (0.00)

9. Other Pre Specified Outcome: Ashworth Spasticity Scale
Time Frame: 3 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Abilhand Questionnaire
Time Frame: 3 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Motor Activity Log
Time Frame: 3 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: fMRI Overactivation in Motor Cortex: Voxel Count and Intensity
Time Frame: 3 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Barthel Index
Description: The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living. Ten variables describing activities of daily living and mobility are scored. The total score ranges 0-100, a higher number being a reflection of greater ability to function independently following hospital discharge.
Time Frame: 3 months
Population: All participants with available data were included. fMRI Control Group no Intervention" subgroup did not have clinical intervention or clinical outcome measures performed, their data was used for the fMRI and TMS component of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | tDCS and no Arm Movement | Sham and no Arm Movement
Number analyzed (Participants) | 7 | 6 | 2 | 1
score on a scale | 66.4 (12.1) | 82.5 (16.0) | 57.5 (10.6) | 50.0 (0.0)

14. Other Pre Specified Outcome: Medical Research Council (MRC) Scale
Description: The muscle scale grades muscle strength on a scale of 0 to 5 in relation to the maximum expected for that muscle. The patient's effort is graded on a scale of 0 (no movement) -5 (muscle contracts normally against full resistance).
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, the entire time of follow-up.
Arm/Group | tDCS and Occupational Therapy | Sham and Occupational Therapy | fMRI Control Group no Intervention | tDCS and no Arm Movement | Sham and no Arm Movement
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/17 | 0/15 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/17 | 0/15 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 9/19 | 3/17 | 0/15 | 2/6 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS and Occupational Therapy (N=19) | Sham and Occupational Therapy (N=17) | fMRI Control Group no Intervention (N=15) | tDCS and no Arm Movement (N=6) | Sham and no Arm Movement (N=4)
recurrent stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient developed bilateral strokes prior to starting therapy, therefore patient was discontinued from study after randomization.
death (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient succumbed to pneumonia two months after completing therapy.
mental status change hospitalisation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient had two episodes of loss of consciousness, no stroke or seizure 1 year after treatment
hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient fell and suffered two successive hip fractures almost a year after treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | tDCS and Occupational Therapy (N=19) | Sham and Occupational Therapy (N=17) | fMRI Control Group no Intervention (N=15) | tDCS and no Arm Movement (N=6) | Sham and no Arm Movement (N=4)
phosphene phenomenon (Nervous system disorders) | 4 | 0 | 0 | 2 | 0 — Resolved with changing the electrode pads. Expected event.
itching or tingtling under the electrode (Product Issues) | 5 | 1 | 0 | 0 | 0 — Expected event, was generally mild and resolved spontaneously within minutes.
vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 — Expected event, resolved spontaneously
sleepiness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 — No treatment was given to this subject, as patient was too sleepy for participation. After 3 consecutive days of inability to perform treatment patient was discontinued from study according to protocol.
car accident (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 — Only bruising, not requiring hospitalisation approx 3 months from treatment.

LIMITATIONS AND CAVEATS:
Slow recruitment and termination before pre-specified number of subjects recruited, attrition due to being lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No